CLINICAL TRIAL: NCT04973514
Title: Perioperative Transfusion Strategies in Adult Congenital Heart Disease Patients Undergoing Cardiac Surgery, Impact on Outcome
Brief Title: Perioperative Transfusion Strategies in Adult Congenital Heart Disease Patients Undergoing Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Denis SCHMARTZ, Anesthesiologists, Head of department, Brugmann University Hospital
Other Study IDs: CHUB_GUCHD
Record Dates: First submitted 2021-04-23; First posted 2021-07-22 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Congenital Heart Disease; Cardiac Surgery; Blood Transfusion; Morbidity, Multiple
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cardiac surgery in grown-up congenital heart disease patients — Analysis of patient blood management, influence on 30 day and 6 month outcome

SUMMARY:
Due to better medical care, a growing number of patients with congenital heart disease reach adulthood. A large number of these patients needs a redo cardiac surgery. No guidelines of best transfusion practice exist for this patient population. A retrospective analysis of all adult patients with congenital heart disease undergoing cardiac surgery between 2000 and 2020 will be performed. Transfusion practices and their influence on outcome at 30 days and 6 month will be evaluated.

DETAILED DESCRIPTION:
Introduction: About 1% of newborns in Belgium have a congenital heart defect. The improvement of intra- and postoperative treatment and the development of new surgical techniques have allowed an increasing management of congenital heart pathologies, making it possible to successfully treat approximately 95% of children with these conditions. The increase in life expectancy of these children has resulted in an ever-increasing proportion of this population reaching adulthood.

Most patients with congenital heart disease, particularly cyanotic conditions, require specialized follow-up in a referral center, given the risk of late complications related to correction or palliation of the primary condition.

Reoperations in adulthood pose a number of challenges for the multidisciplinary team managing these patients: more complex surgical approach (adhesions, altered in situ anatomy, development of collateral circulation, persistence of intra- or extra-cardiac shunts...). The operative risk but also the infectious risk are clearly increased in this population.

The risk of bleeding, which is already high in cardiac surgery, particularly due to the use of extracorporeal circulation, is also increased by the re-intervention itself. This is potentially accompanied by greater exposure to allogeneic blood products, which has been associated with increased postoperative morbidity and mortality.

Various techniques have been developed to reduce the risk of bleeding in cardiac surgery, including the use of anti-fibrinolytic agents, avoidance of deep hypothermia, reduction of vascular filling to avoid excessive hemodilution, and application of a permissive hypotension and restrictive transfusion strategy. The ultimate goal of integrating these techniques into our transfusion practices is to improve patient outcomes by reducing exposure to blood products. There are currently no recommendations on good transfusion practices for the management of these patients with congenital heart disease who require cardiac re-intervention in adulthood. There are also few studies specific to this population in the current literature.

Objectives: The main objective of the study is to analyze, in our center, if the transfusion practices (measures to decrease the risk of bleeding, transfusion of red blood cells (RBCs) and/or blood derivatives), in patients who have had a re-intervention of congenital heart surgery, are determinant to reduce morbidity and mortality in the following 30 days and 6 months Type of study and design: Retrospective and descriptive study by extraction of patients who underwent cardiac surgery, at the Brugmann University Hospital, between the year 2000 to the year 2020, by analysis of the medical charts.

Patients: Grown-up congenital heart disease patients re-operated from cardiac surgery between January 2000 to December 2020.

Inclusion criteria: All patients with congenital heart disease reoperated from a new cardiac surgery under extracorporeal circulation, at Brugmann University Hospital, between the year 2000 to the year 2020.

Exclusion criteria: Patients with cardiac surgery without cardiopulmonary bypass, patients with acquired heart disease, patients who had a re-intervention due to a complication within 30 days postoperatively.

Statistical evaluation: Descriptive analyses will be used and further analyses will be performed based on preliminary results and hypotheses raised. The patients' data will be put in an anonymized file and analyzed later.

Variables to be collected: demographic data; type of procedure; personal history of the patient; clinical symptomatology; pre-op, intra-op and post-op treatment; complementary pre-, per-, and post-op examinations (radiological, laboratories), operative data (surgical procedure performed, blood loss, blood component transfusion (red blood cells, platelets, plasma), fluid balance, use of anti-fibrinolytics) ; hemodynamic monitoring (intraoperative vital parameters), duration of cardiopulmonary bypasss (CPB) time, aortic clamping time, intraoperative and postoperative complications, death, length of stay in intensive care and total length of stay.

ELIGIBILITY:
Inclusion Criteria:

* All adult congenital heart disease patients undergoing cardiac surgery with cardiopulmonary bypass between 2000 and 2020 at Brugmann University Hospital

Exclusion Criteria:

* Off-pump cardiac surgery
* re-intervention within 30 days of cardiac surgery due to complications

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All adult congenital heart disease patients undergoing cardiac surgery with cardiopulmonary bypass between 2000 and 2020 at Brugmann University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-07-20 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Outcome 30 day | 30 days
  Outcome at 30 days postoperative, defined as new organ failure or death
Outcome 6 months | 6 month
  Outcome at 6 months postoperatively, defined as new organ failure or death

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miltner B, Pierard L, Seghaye MC. [Follow up of adults with congenital heart disease]. Rev Med Liege. 2012 Jul-Aug;67(7-8):407-12. French. PMID 22984760
- [Background] Webb GD. Care of adults with congenital heart disease--a challenge for the new millennium. Thorac Cardiovasc Surg. 2001 Feb;49(1):30-4. doi: 10.1055/s-2001-9918. PMID 11243519
- [Background] Dore A, Glancy DL, Stone S, Menashe VD, Somerville J. Cardiac surgery for grown-up congenital heart patients: survey of 307 consecutive operations from 1991 to 1994. Am J Cardiol. 1997 Oct 1;80(7):906-13. doi: 10.1016/s0002-9149(97)00544-4. PMID 9382007
- [Background] Rychik J, Atz AM, Celermajer DS, Deal BJ, Gatzoulis MA, Gewillig MH, Hsia TY, Hsu DT, Kovacs AH, McCrindle BW, Newburger JW, Pike NA, Rodefeld M, Rosenthal DN, Schumacher KR, Marino BS, Stout K, Veldtman G, Younoszai AK, d'Udekem Y; American Heart Association Council on Cardiovascular Disease in the Young and Council on Cardiovascular and Stroke Nursing. Evaluation and Management of the Child and Adult With Fontan Circulation: A Scientific Statement From the American Heart Association. Circulation. 2019 Aug 6;140(6):e234-e284. doi: 10.1161/CIR.0000000000000696. Epub 2019 Jul 1. PMID 31256636
- [Background] Haapanen H, Tsang V, Kempny A, Neijenhuis R, Kennedy F, Cullen S, Walker F, Kostolny M, Hsia TY, Van Doorn C. Grown-up Congenital Heart Surgery in 1093 Consecutive Cases: A "Hidden" Burden of Early Outcome. Ann Thorac Surg. 2020 Nov;110(5):1667-1676. doi: 10.1016/j.athoracsur.2020.01.071. Epub 2020 Mar 5. PMID 32147413
- [Background] Talwar S, Kumar MV, Sreenivas V, Choudhary SK, Sahu M, Airan B. Factors determining outcomes in grown up patients operated for congenital heart diseases. Ann Pediatr Cardiol. 2016 Sep-Dec;9(3):222-8. doi: 10.4103/0974-2069.189113. PMID 27625519
- [Background] Berdat PA, Immer F, Pfammatter JP, Carrel T. Reoperations in adults with congenital heart disease: analysis of early outcome. Int J Cardiol. 2004 Feb;93(2-3):239-45. doi: 10.1016/j.ijcard.2003.04.005. PMID 14975553
- [Background] Vida VL, Berggren H, Brawn WJ, Daenen W, Di Carlo D, Di Donato R, Lindberg HL, Corno AF, Fragata J, Elliott MJ, Hraska V, Kiraly L, Lacour-Gayet F, Maruszewski B, Rubay J, Sairanen H, Sarris G, Urban A, Van Doorn C, Ziemer G, Stellin G. Risk of surgery for congenital heart disease in the adult: a multicentered European study. Ann Thorac Surg. 2007 Jan;83(1):161-8. doi: 10.1016/j.athoracsur.2006.07.045. PMID 17184653
- [Background] Brevig J, McDonald J, Zelinka ES, Gallagher T, Jin R, Grunkemeier GL. Blood transfusion reduction in cardiac surgery: multidisciplinary approach at a community hospital. Ann Thorac Surg. 2009 Feb;87(2):532-9. doi: 10.1016/j.athoracsur.2008.10.044. PMID 19161774
- [Background] Kuduvalli M, Oo AY, Newall N, Grayson AD, Jackson M, Desmond MJ, Fabri BM, Rashid A. Effect of peri-operative red blood cell transfusion on 30-day and 1-year mortality following coronary artery bypass surgery. Eur J Cardiothorac Surg. 2005 Apr;27(4):592-8. doi: 10.1016/j.ejcts.2005.01.030. PMID 15784356
- [Background] Wilkinson KL, Brunskill SJ, Doree C, Trivella M, Gill R, Murphy MF. Red cell transfusion management for patients undergoing cardiac surgery for congenital heart disease. Cochrane Database Syst Rev. 2014 Feb 7;2014(2):CD009752. doi: 10.1002/14651858.CD009752.pub2. PMID 24510598
- [Background] Giamberti A, Chessa M, Abella R, Butera G, Carlucci C, Nuri H, Frigiola A, Ranucci M. Morbidity and mortality risk factors in adults with congenital heart disease undergoing cardiac reoperations. Ann Thorac Surg. 2009 Oct;88(4):1284-9. doi: 10.1016/j.athoracsur.2009.05.060. PMID 19766822